CLINICAL TRIAL: NCT02533973
Title: Long-term Treatment of Scalp Psoriasis With Xamiol® Gel in a Large Adult Chinese Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0076-1079
Record Dates: First submitted 2015-08-20; First posted 2015-08-27 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2018-11

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xamiol® gel (Active Comparator): calcipotriol 50mcg/g plus betamethasone 0.5 mg/g (as diproprionate) once daily as required, for up to 28 weeks
  Interventions: Drug: Xamiol® gel
- . Daivonex® scalp solution (Active Comparator): calcipotriol 50mcg/g twice daily as required, for up to 28 weeks
  Interventions: Drug: Daivonex® scalp solution

INTERVENTIONS:
Drug: Xamiol® gel
  Arms: Xamiol® gel
Drug: Daivonex® scalp solution
  Arms: . Daivonex® scalp solution

SUMMARY:
A phase 4 trial comparing the safety and efficacy of treatment with Xamiol® gel (calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate)) once daily (as required) with Daivonex® scalp solution (calcipotriol 50 mcg/g) twice daily (as required) in Chinese subjects with scalp psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent has been obtained.
2. Subjects of either gender 18 years of age or above.
3. At visit 1, a clinical diagnosis of scalp psoriasis which is:

   * of an investigator's assessment of clinical signs of the scalp of at least ≥ 2 in one of the clinical signs, redness, thickness, and scaliness, and at least 1 in each of the other two clinical signs, and total score ≥ 4
   * of an extent of 10% or more of the total scalp area
   * of at least mild severity according the investigator's global assessment
4. Clinical signs of psoriasis vulgaris on trunk and/or limbs, or subject earlier diagnosed with psoriasis vulgaris on trunk and/or limbs.
5. Female of childbearing potential using a reliable method of contraception for at least 1 month before the trial start and during the course of the trial (e.g., oral contraceptive pill, intrauterine device, contraceptive patches, implantable contraception, condoms) or females of non-childbearing potential (i.e. postmenopausal (absence of menstrual bleeding for 2 years), hysterectomy, bilateral ovariectomy, or tubal section/ligation).

Exclusion Criteria:

1. Current diagnosis of guttate, erythrodermic, exfoliative, or pustular psoriasis.
2. Subjects with any of the following conditions present on the scalp area: viral lesions, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, acne rosacea, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers, and wounds.
3. Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation and during the trial:

   * etanercept (Yisaipu) - within 4 weeks prior to randomisation
   * infliximab (Remicade) - within 2 months prior to randomisation
   * other products: within 4 weeks/5 half-lives (whichever is longer) prior to randomisation
4. Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, methotrexate, ciclosporin and other immunosuppressant's, TCM [(traditional Chinese Medicine)]) within 4 weeks prior to randomisation or during the trial.
5. PUVA therapy within 4 weeks prior to randomisation or during the trial.
6. UVB therapy within 2 weeks prior to randomisation or during the trial.
7. Therapies within 2 weeks prior to randomisation and during the trial:

   * Topical treatment of body psoriasis with very potent (WHO group IV) corticosteroids
   * Topical treatment of face psoriasis with potent or very potent (WHO group III and IV) corticosteroids
   * Any topical treatment of the scalp (except for non-steroid medicated shampoos and emollients)
8. Known or suspected renal insufficiency or hepatic disorders or severe heart disease.
9. Clinical signs or symptoms of Cushing's disease or Addison's disease.
10. Known or suspected hypersensitivity to component(s) of IMPs
11. Current participation in any other interventional clinical trial
12. Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within 4 weeks/5 half-lives (whichever is longer) prior to randomisation.
13. Previously participated in a clinical trial within 4 weeks prior to randomisation.
14. In the opinion of the (sub) investigator, the subject is unlikely to comply with the clinical trial protocol (e.g. due to alcoholism, drug addiction or psychotic state).
15. Females who are pregnant, or of child-bearing potential and wish to become pregnant during the trial, or who are breast-feeding.
16. Females of child-bearing potential with a positive urine pregnancy test at visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
safety of Xamiol® gel (adverse events) | 28 Weeks
  To establish the safety of Xamiol® gel over a long period for up to 28 weeks of treatment in Chinese subjects. Incidence of adverse drug reactions of any type and Incidence of adverse events of concern associated with long-term corticosteroid use on the scalp.

SECONDARY OUTCOMES:
Efficacy of Xamiol® gel ( percentage of visits in which subjects had "Treatment success" according to Investigator's Global Assessment) | 28 Weeks
  To establish the efficacy of Xamiol® gel over a long period for up to 28 weeks of treatment in Chinese subjects. The percentage of visits in which subjects had "Treatment success" according to Investigator's Global Assessment of disease severity during the treatment. The percentage of visits in which subjects had "Treatment success" according to subject's global assessment of disease severity during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, MD, PHD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No